CLINICAL TRIAL: NCT06690320
Title: Effect of Planned Education on Health Beliefs and Fatalism in Women at High Risk of Breast Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gülsen Calıs, NURSE, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 23-4.1T/56
Record Dates: First submitted 2024-10-20; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Health Behavior; Breast Self-Examination
Keywords: breast cancer; health belief model; fatalism; public health nursing; nurse; early diagnosis of cancer
MeSH Terms: conditions — Breast Neoplasms; Health Behavior; Breast Self-Examination

STUDY DESIGN:
Intervention Model Description: Research population: The population of this research consists of women who received 301 or more points from the breast cancer risk assessment form who applied to the family medicine polyclinic and general surgery breast polyclinic of Ordu University Training and Research Hospital in Ordu province between 2023-2024.
  In the study, the sample size was calculated at a 95% confidence level using the "G. Power-3.1.9.2" program. As a result of the analysis, the standardized effect size was found to be 1.1270 at the α=0.05 level, based on the previous study, and the minimum sample size was calculated as 60 with a theoretical power of 0.99, 30 for the experimental group and 30 for the control group. Considering the losses, it was decided to collect 20% more and it was aimed to reach 72 people, 36 for the experimental group and 36 for the control group.
Who Masked: Outcomes Assessor
Masking Description: statistical evaluation of the research results will be made by an expert other than the researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No application will be made to the control group. After the research is completed, a planned training program can be applied to the experimental group upon request by the researcher within the framework of ethical responsibilities.
- experiment group (Experimental): A one-session planned training program will be applied to the experimental group.
  Interventions: Behavioral: IMPLEMENTATION OF A PLANNED EDUCATION PROGRAM ON HEALTH BELIEF MODEL AND FATUALIST TENDENCIES IN WOMEN AT HIGH RISK OF BREAST CANCER

INTERVENTIONS:
Behavioral: IMPLEMENTATION OF A PLANNED EDUCATION PROGRAM ON HEALTH BELIEF MODEL AND FATUALIST TENDENCIES IN WOMEN AT HIGH RISK OF BREAST CANCER — Description: By examining the parameters of the health belief model and fatalism scales, 6 targets were determined for these scale parameters. The targets were prepared to gain early diagnosis behaviors in breast cancer. By using the breast model, the behavior will be demonstrated in practice
  Arms: experiment group

SUMMARY:
Purpose: This project aims to examine the effects of planned education on health beliefs and fatalism in women at high risk of breast cancer. When national and international literature was examined, no project was found in which the health beliefs and fatalism of high-risk women in breast cancer were determined and then the results were evaluated by implementing a planned education. Therefore, planning an original project in this field aims to contribute to the literature.

Scope and Target Group: The project will be carried out with women who applied to Ordu Education and Research Hospital Family Medicine and General Surgery Breast Polyclinic within the borders of Ordu province and who received 301 and above points from the breast cancer risk assessment form (N=72). Ordu University Education and Research Hospital is a hospital that provides services with an affiliation protocol within the framework of the "Regulation on the Methods and Principles of Cooperation with the Joint Use of the Institutions and Organizations of the Ministry of Health and its Affiliated Organizations and the Relevant Units of State Universities".

Method and Expected Result: The project was planned as a randomized controlled experimental follow-up study with a pre-test-post-test control group design in order to examine the effect of planned education on health beliefs and fatalism in women at high risk of breast cancer. Planned education intervention will be applied to women at high risk of breast cancer whose health beliefs and fatalistic tendencies have been determined. Planned education will provide breast self-examination (BSE) on the model closest to human tissue, and pathologies related to breast cancer will be detected on the model by touching the model. An approach based on raising awareness of breast cancer and learning early diagnosis methods through doing and living experience will be provided. Therefore, it is expected that the planned education applied by doing and experiencing on a model close to human tissue will be effective in gaining and implementing health behaviors in women with known health beliefs and fatalistic tendencies at high risk of breast cancer. In addition, it is expected that the application by doing and experiencing will be effective in gaining permanent health behaviors.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer in women, accounting for approximately 12% of cancer cases. According to the World Health Organization, 2.3 million women were diagnosed with breast cancer in 2020, and 685,000 people lost their lives. Breast cancer ranks second in cancer death statistics in Turkey. Approximately 15,000 women are diagnosed with breast cancer every year. The incidence is highest in the 25-49 age group with 35.6%.The increase in breast cancer prevalence rates in the world and in Turkey and the decreasing age of onset show how important it is to increase public awareness of this issue and their participation in screening programs. Today, 30-50% of cancer can be prevented. This can be achieved by avoiding risk factors and implementing existing evidence-based prevention strategies. Some of the prevention strategies are; reaching women at risk for breast cancer, early diagnosis, and providing health behaviors through education.

The American Cancer Society states that there are women at high risk for breast cancer, and that factors such as gender, age, history, family history, early menarche, etc. that increase the risk factor should be evaluated In this context, it is necessary to evaluate breast cancer risk status correctly. Models aimed at predicting the risk of developing cancer are useful for implementing prevention strategies such as planning education and providing counseling In Turkey, the 'Breast Cancer Risk Assessment Form' is used for calculations aimed at predicting the risk of developing breast cancer. Thus, the risk status in breast cancer can be determined and early precautions can be taken according to the situation. Early stage diagnosis in breast cancer provides a good prognosis and is of critical importance for long-term survival. In this project, reaching high-risk women in breast cancer using the 'Breast Cancer Risk Assessment Form' and calculating their risk levels is seen as an important gain.

The probability of recovery is high for many early-diagnosed cancers. Especially considering that the age at which breast cancer screening begins varies among high-risk women, reaching these high-risk women at the right time in society, ensuring that individual risk is calculated and perceived correctly, is important for gaining health behaviors appropriate for early diagnosis methods. In this direction; It is necessary to gain health behaviors such as early diagnosis methods such as breast self-examination (BSE), clinical breast examination (CBE) and mammography to high-risk women in breast cancer through planned education. Another gain of this project is to gain health behaviors in early diagnosis in breast cancer through planned education.

Global Breast Cancer Initiative (GBCI); recommends disseminating early diagnosis methods and creating breast cancer awareness for health promotion and development Awareness can only be achieved through educational activities carried out within the framework of a developed plan. It is stated that women have information needs (treatment, breast cancer symptoms and breast self-examination) and support needs (learning to do BSE, women's concerns for themselves and their relatives, having professional breast examination at the health institution) in breast cancer prevention. In this context, the importance of planned education is increasing in order to provide information and support needs in breast cancer prevention. The importance of providing planned education to women is also emphasized in many studies. The selection of the method in the planned education should be in a way that will meet the information and support needs. Especially BSE; It becomes more permanent when it provides experience-based learning through 'doing, living' on a breast model. In this project, especially with a planned education based on 'doing, living' experience-based learning, providing women at high risk of breast cancer with the experience of feeling and finding breast cancer signs and symptoms on a 'breast model', experiencing pathological formations and performing BSE examination skills with steps, and ensuring the permanence of health behavior is seen as an important gain.

On the other hand, it is stated that the health belief status and fatalism approach of the individual are also important for the early diagnosis behaviors of breast cancer to be permanent. These health beliefs can be preventive or supportive in some cases. Fatalism and health belief are important predictors in the potential emergence of the behavior.Therefore, knowing and measuring the health belief and fatalism status of women is important for women at high risk of breast cancer. Another output of the project is the measurement of the health beliefs and fatalism status of women at high risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

• Being 30 years of age or older, Being at least literate, Getting a score of 301 or higher from the Breast Cancer Risk Assessment Form, Not having vision or hearing loss that would prevent communication, Accepting participation in the study voluntarily.

Exclusion Criteria:

* Being a healthcare professional,

  * Having received genetic counseling for breast cancer due to a breast cancer diagnosis in a 1st, 2nd or 3rd degree relative,
  * Having received breast cancer early diagnosis training within the last 1 year,
  * Those who were diagnosed with breast cancer and received treatment during the study period will not be included in the study

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Champion's Health Belief Model Scale | 15 days
  The health belief model scale will be applied to the experimental and control groups. Pre-test-post-test data to evaluate the effectiveness of the intervention for nurses who will attempt to change/improve women's beliefs and behaviors regarding breast cancer and screening behaviors. In the Turkish adaptation of the scale. CSİMO has 6 sub-dimensions and the items are listed in the order of the data below. Each sub-dimension of the scale is evaluated separately, the total score including the entire scale is not calculated. Women who score low on the "perception of obstacle" sub-scale and high on other sub-scales show that they have positive attitudes and beliefs

SECONDARY OUTCOMES:
Powe's Breast Cancer Fatalism Scale | 15 days
  Powe's Breast Cancer Fatalism Scale will be applied to the experimental and control groups. The scale consists of 11 items. It is answered as yes / no. A "yes" answer is calculated as 1 point, a "no" answer is calculated as 0 points.

OTHER OUTCOMES:
BREAST CANCER RISK ASSESSMENT FORM | Baseline
  This is the form used by people receiving the service in the National Family Planning Service Guide (2005) to determine the risk of women from breast cancer. The form was also developed by the American Cancer Society and is recommended for use by the Ministry of Health in Turkey. The Breast Cancer Risk Assessment Form consists of six sections and 20 items. Women who receive 301 and above from this form are included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: gülşen çalış, Principal Investigator — gulsencalis81@gmail.com
Locations (1):
- Ege UnIversty, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andic S, Karayurt O. Determination of information and support needs of first degree relatives of women with breast cancer. Asian Pac J Cancer Prev. 2012;13(9):4491-9. doi: 10.7314/apjcp.2012.13.9.4491. PMID 23167367
- [Result] Kharameh ZT, Foroozanfar S, Zamanian H. Psychometric properties of the Persian version of Champion's Health Belief Model Scale for colorectal cancer screening. Asian Pac J Cancer Prev. 2014;15(11):4595-9. doi: 10.7314/apjcp.2014.15.11.4595. PMID 24969891
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: world healt organization — https://www.who.int/data/gho/data/themes/mortality-and-global-health-estimates/ghe-leading-causes-of-death
- See also: T.C. SAĞLIK BAKANLIĞI HALK SAĞLIĞI GENEL MÜDÜRLÜĞÜ — https://hsgm.saglik.gov.tr/tr/